CLINICAL TRIAL: NCT05928377
Title: Patient Perspectives in Testicular Cancer Clinical Trials: Insights Into Participating in Studies for Testicular Cancer
Brief Title: Unveiling Patient Experiences in Testicular Cancer Clinical Trials
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 80505443
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Testicular Cancer
Keywords: testicular cancer
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical research participation has historically been heavily biased toward specific demographics.

Several people will be invited to enroll in this study so that it may collect a variety of data about testicular cancer clinical study experiences and identify barriers to participation as well as the causes of participants' failure or withdrawal.

People with testicular cancer who are invited to take part in medical research will benefit from the analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Diagnosis of testicular cancer
* No prior treatment for testicular cancer

Exclusion Criteria:

* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Enrolled in another research study
* Inability to provide written informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Testicular cancer patients who are actively considering enrolling in a clinical trial for the said condition, but have not yet completed enrollment and randomization phases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of testicular cancer patients who decide to enroll in a clinical trial | 3 months
Rate of testicular cancer patients who remain in a clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ljungman L, Eriksson LE, Flynn KE, Gorman JR, Stahl O, Weinfurt K, Wiklander M, Lampic C, Wettergren L. Sexual Dysfunction and Reproductive Concerns in Young Men Diagnosed With Testicular Cancer: An Observational Study. J Sex Med. 2019 Jul;16(7):1049-1059. doi: 10.1016/j.jsxm.2019.05.005. PMID 31255211
- [Background] Selvi I, Sarikaya S, Basar H. Is testicular microlithiasis a really innocent condition? Its effects on oncological outcomes of germ cell testicular cancer: An observational study. Arch Esp Urol. 2020 Apr;73(3):215-229. English, Spanish. PMID 32240112
- [Background] Pedersen MR, Sloth Osther PJ, Nissen HD, Vedsted P, Moller H, Rafaelsen SR. Elastography and diffusion-weighted MRI in patients with testicular microlithiasis, normal testicular tissue, and testicular cancer: an observational study. Acta Radiol. 2019 Apr;60(4):535-541. doi: 10.1177/0284185118786063. Epub 2018 Jul 3. PMID 29969051